CLINICAL TRIAL: NCT04436926
Title: The Neural Basis of Approach Bias Modification in Opioid Users With Chronic Pain
Brief Title: Opioid Approach Bias Modification
Acronym: OABM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-29607
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Opioid Use; Chronic Pain
Keywords: opioid; approach bias; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid approach bias training (Experimental): Immediately following screening, patients will be randomly assigned to receive 6 sessions of opioid approach bias modification taking place over two weeks.
  Interventions: Behavioral: opioid approach bias modification
- sham training (Sham Comparator): Immediately following screening, patients will be randomly assigned to receive 6 sessions of sham training taking place over two weeks.
  Interventions: Behavioral: sham training

INTERVENTIONS:
Behavioral: opioid approach bias modification — The investigators will use a training version of the Approach-Avoidance Task (AAT), in which patients are asked to respond to the format of presented pictures, irrespective of the pictures' content. Pushing a presented picture away will decrease picture size, whereas pulling a picture closer will increase size. There are 2 categories of pictures; 20 different opioid and 20 different non-medication alternative pain managing activities. Training effect is achieved by presenting opioid pictures in push format only and non-opioid pictures in pull format only. Two hundred training trials are presented per session.
  Arms: opioid approach bias training
Behavioral: sham training — Sham training is identical to opioid approach bias training, except pictures are presented randomly in both formats.
  Arms: sham training

SUMMARY:
To investigate the neurobiological mechanisms underlying opioid approach bias during a pilot RCT of opioid approach bias modification. The investigators are combining novel ultra-high field MRI technology with the promising treatment of modifying cognitive bias away from detrimental prescription drug use will generate novel neural data and potentially yield a new therapeutic tool to reduce problematic opioid use.

DETAILED DESCRIPTION:
The proposed study is a pilot prospective, parallel groups, randomized, double blind, sham training-controlled, 6-session (over 2 weeks) clinical trial of opioid approach bias modification (OABM) in 20 male and female veterans with chronic pain at high risk for opioid-related adverse events at the San Francisco Veterans Affairs Health Care System, between ages 18-69. The study consists of screening, 2-week cognitive training, Week-3 post-assessment. Assessment of the neurobiological mechanisms of opioid approach bias will be administered at baseline and Week-3.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veterans eligible for VA services
* Ages 18-69
* Chronic pain (current pain lasting ≥ 90 days)
* Prescribed chronic opioids (≥ 90 days in past year)
* High risk for opioid-related averse outcomes (≥ 20mg morphine equivalent daily dose).

Exclusion Criteria:

* Psychotic, bipolar disorders or other psychiatric disorders judged to be unstable by the PI
* Current or past history of the following: intrinsic cerebral tumors, cerebrovascular accident/disease, brain aneurysm, arteriovenous malformations, surgical implantation of neurostimulators or cardiac pacemakers, demyelinating and neurodegenerative diseases, penetrating traumatic brain injury, and any other MRI contraindications.
* No female participant will be pregnant or actively attempting to conceive to prevent any unnecessary exposure to high magnetic fields or radio frequency energy to the unborn child.
* Concurrent participation in a treatment study
* Moderately Severe/Severe withdrawal from opioids based on a score of 25 or more on the Clinical Opiate Withdrawal Scale (COWS)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in reaction time on an opioid approach-avoidance task across time, baseline to end of treatment, week 3 | baseline to end of treatment, week 3
  millisecond reaction time of (opioid push - opioid pull) - (non-opioid push - opioid pull) on an opioid approach-avoidance task where participants are asked to respond to the format of presented pictures, irregardless of the content. There are two categories of pictures; 20 different opioid pictures and 20 different non-opioid pictures, with two-hundred trials. Millisecond reaction time will be measured at baseline, prior to each training session during the 2-week training period, and at week 3 post training assessment. Primary outcome is change in reaction time across time in active vs. sham condition.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Batki, MD, Principal Investigator — University of California, San Francisco; David Pennington, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- VA Medical Center San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No